CLINICAL TRIAL: NCT06228131
Title: Detection of hCG in Early Pregnancy Clinical Samples
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IHC-3000-LCFA02
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Early Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples Without DNA — urine sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects who provided early pregnancy urine samples

SUMMARY:
To evaluate the detection of hCG in the early pregnancy urine samples by Human chorionic gonadotropin (HCG) test system.

ELIGIBILITY:
Inclusion Criteria:

* Female；
* 18-55 years of age；
* In a state of preparing for pregnancy;
* Voluntary and sign informed consent form.

Exclusion Criteria:

* Within 8 weeks of childbirth or abortion；
* The investigator has reason to believe that it is inappropriate for subjects to participate in the study.

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: There were 241 subjects who planned to conceive but did not conceive participating in the clinical trial. Of these, 73 women successfully conceived and provided a full cycle of urine samples(10 days, from day -8 to day +1 relative to the expected period) .
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the detection of hCG in the early pregnancy urine samples by investigational device. | 10day
  Percentage Pregnancy Results (%) for early pregnancy urine samples on different days from day -8 to day +1 relative to the expected period.
  Percentage Pregnancy Results (%): 79% (day -5 relative to the expected period)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Teaching hospital of Tianjin University of Traditional Chinese Medicine, Tianjin
  - Internet Hospital of Tianjin Medical University General Hospital, Tianjin